CLINICAL TRIAL: NCT00849082
Title: Phase III Randomized Comparison of Pelvic Radiotherapy Alone vs Pelvic Radiotherapy Plus the LHRH Analogue Goserelin and Cyproterone Acetate in Carcinoma of the Prostate at High Risk for Metastasis
Brief Title: Radiation Therapy With or Without Goserelin and Cyproterone in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-22863; EORTC-22863
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyproterone Acetate; Goserelin; Radiotherapy

INTERVENTIONS:
Drug: cyproterone acetate
Drug: goserelin acetate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high energy x rays to kill tumor cells. This may be an effective treatment for prostate cancer. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as goserelin and cyproterone, may lessen the amount of androgens made by the body and reduces the amount of androgens available to the body. It is not yet know whether radiation therapy alone is more effective than radiation therapy given together with goserelin and cyproterone in treating patients with prostate cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared to giving radiation therapy together with goserelin and cyproterone in treating patients with prostate cancer that is at high risk for metastasis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the ability of adjuvant hormone therapy with an LHRH agonist (Goserelin depot) to produce an increased disease-free survival and to prolong overall survival when initiated during the first week of radiotherapy in prostatic cancer patients with a high risk of developing metastatic disease.

OUTLINE: Randomized study. Arm I: Radiotherapy. Whole-pelvic irradiation using photons with a recommended energy of at least 10 MV (Co60 therapy is acceptable if higher energy unavailable). Arm II: Radiotherapy plus 2-Drug Combination Hormonal Therapy. Whole-pelvic irradiation as in Arm I; plus Goserelin, ZDX, NSC-606864; Cyproterone acetate, CPTR, NSC-81430.

PROJECTED ACCRUAL: 400 patients will be entered over 5 years. At least 75 patients on each arm should be followed until relapse.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven prostatic adenocarcinoma of the following TNM stages and WHO grades: T1 or T2 and grade G3 T3 or T4 and any histologic grade No evidence of distant metastases No evidence of positive common iliac or para-aortic lymph nodes Confirmed by bone scan, chest x-ray, negative ultrasound or CT of the liver, and CT of the retroperitoneum and/or bipedal lymphangiography Extraperitoneal pelvic lymph node biopsy may be either positive or negative provided stage and grade criteria are met

PATIENT CHARACTERISTICS: Age: Under 80 Performance status: WHO 0-2 Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No history of second malignancy except basal cell skin carcinoma

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for prostate cancer Endocrine therapy: No prior hormonal therapy for prostate cancer Radiotherapy: No prior radiotherapy for prostate cancer Surgery: No prior radical prostatectomy No prior transperitoneal lymph node staging

Max Age: 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1987-05; Primary Completion 1995-11 (Actual)

PRIMARY OUTCOMES:
Disease-free survival
Survival
Toxicity/morbidity of treatment,
Locoregional remission rate
Time to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bolla, MD, Study Chair — CHU de Grenoble - Hopital de la Tronche

REFERENCES:
- [Result] Bolla M, Van Tienhoven G, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Billiet I, Torecilla JL, Pfeffer R, Cutajar CL, Van der Kwast T, Collette L. External irradiation with or without long-term androgen suppression for prostate cancer with high metastatic risk: 10-year results of an EORTC randomised study. Lancet Oncol. 2010 Nov;11(11):1066-73. doi: 10.1016/S1470-2045(10)70223-0. Epub 2010 Oct 7. PMID 20933466
- [Result] Ataman F, Zurlo A, Artignan X, van Tienhoven G, Blank LE, Warde P, Dubois JB, Jeanneret W, Keuppens F, Bernier J, Kuten A, Collette L, Pierart M, Bolla M. Late toxicity following conventional radiotherapy for prostate cancer: analysis of the EORTC trial 22863. Eur J Cancer. 2004 Jul;40(11):1674-81. doi: 10.1016/j.ejca.2003.12.027. PMID 15251156
- [Result] Bolla M, Collette L, Blank L, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Mattelaer J, Lopez Torecilla J, Pfeffer JR, Lino Cutajar C, Zurlo A, Pierart M. Long-term results with immediate androgen suppression and external irradiation in patients with locally advanced prostate cancer (an EORTC study): a phase III randomised trial. Lancet. 2002 Jul 13;360(9327):103-6. doi: 10.1016/s0140-6736(02)09408-4. PMID 12126818
- [Result] Zurlo A, Collette L, van Tienhoven G, Blank L, Warde P, Dubois J, Jeanneret W, Storme G, Bernier J, Kuten A, Pierart M, Bolla M; EORTC Radiotherapy and Genito-Urinary Tract Cancer Groups. Acute toxicity of conventional radiation therapy for high-risk prostate cancer in EORTC trial 22863. Eur Urol. 2002 Aug;42(2):125-32. doi: 10.1016/s0302-2838(02)00257-9. PMID 12160582
- [Result] Bolla M, Gonzalez D, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Gil T, Collette L, Pierart M. Improved survival in patients with locally advanced prostate cancer treated with radiotherapy and goserelin. N Engl J Med. 1997 Jul 31;337(5):295-300. doi: 10.1056/NEJM199707313370502. PMID 9233866
- [Result] Dusserre A, Garavaglia G, Giraud JY, Bolla M. Quality assurance of the EORTC radiotherapy trial 22863 for prostatic cancer: the dummy run. Radiother Oncol. 1995 Sep;36(3):229-34. doi: 10.1016/0167-8140(95)01612-k. PMID 8532911